CLINICAL TRIAL: NCT04683328
Title: An Adaptive, Randomized, Double-blinded, Placebo-controlled, Phase II/III Trial of Monoclonal Antibody SCTA01 Against SARS-CoV-2 in Patients With Severe COVID-19 Admitted to High Dependence or Intensive Care Unit (MASP3 Trial)
Brief Title: The Safety and Efficacy of SCTA01 Against COVID-19 in Patients Admitted to High Dependence or Intensive Care
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCTA01-C301
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — upanovimab

STUDY DESIGN:
Intervention Model Description: SCTA01+BSC vs Placebo+BSC
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCTA01 Group (Experimental): SCTA01+Best Supportive Care
  Interventions: Biological: SCTA01
- Placebo Group (Placebo Comparator): Placebo+Best Supportive Care
  Interventions: Biological: SCTA01 Placebo

INTERVENTIONS:
Biological: SCTA01 — Recombinant anti-SARS-CoV-2 spike protein monoclonal antibody
  Arms: SCTA01 Group
Biological: SCTA01 Placebo — The excipients of SCTA01
  Arms: Placebo Group

SUMMARY:
This is an adaptive, randomized, double-blinded, placebo-controlled, Phase II/III study conducted to evaluate the effect of SCTA01 on participant survival and clinical efficacy in participants with severe COVID-19 admitted to high dependence or ICUs.

The study duration of subject participation will be up to: 120 days Participants will receive a single intravenous (IV) infusion of SCTA01 at Treatment day 1. Follow up visits will be up to 120 days or early withdrawal visit.

DETAILED DESCRIPTION:
The study is a multicenter, adaptive, randomized, double-blinded, and placebo-controlled Phase II/III trial. It will be conducted globally. The study will evaluate the efficacy and safety of SCTA01 compared to placebo both given with BSC in participants with severe COVID-19. The subjects will be randomized by 1:1 ratio to SCTA01 and placebo group. The primary objective of the study is to evaluate participant survival from randomization to Day 29 between study group and control group. At the end of the Phase II part of the study, an interim analysis will be performed for safety run-in and futility stopping.

ELIGIBILITY:
Inclusion Criteria:

* Male and female of ≥18years at time of enrollment;
* Subject (or legally authorized representative [LAR]) is able and willing to provide written or verbal informed consent, which includes compliance with study requirements and restrictions listed in the consent form.
* Female subjects must agree to use an approved highly effective birth control (BC) method (<1% failure rate per year) throughout the study (until completion of the Day 85 Follow-up Visit), unless documented to have a reproductive status of non-childbearing potential or is postmenopausal:

  1. Non-childbearing potential defined as pre-menopausal female with medical history of bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries), or hysterectomy; hysteroscopic sterilization,
  2. Postmenopausal defined as 12 months of spontaneous amenorrhea
* Woman of childbearing potential (WCBP) who is already using an established method of highly effective contraception or agrees to use one of the allowed BC methods listed in the protocol, for at least 28 days prior to the start of dosing (as determined by the Investigator or designee) to sufficiently minimize the risk of pregnancy throughout study participation (until completion of the Day 90 Follow-up Visit).
* Hospitalized participants with severe COVID-19（6-8 point on WHO 10-Point Ordinal Scale):

  1. Point 6: Oxygen by NIV or high flow;
  2. Point 7: Intubation and MV, pO2/FiO2 ≥ 150 mmHg or SpO2/FiO2 ≥ 200 mmHg;
  3. Point 8: MV pO2/FiO2 < 150 mmHg (or SpO2/FiO2 < 200 mmHg) or vasopressors .
* Biological samples (not limited to any specific type) collected within 72 hours (allow retesting for potential subjects that tested positive beyond 72 hours) before randomization is laboratory-confirmed as SARS-CoV-2 infection (PCR, etc.);
* ≤ 14 days since the onset of COVID-19 symptoms.

Exclusion Criteria:

* Subject has been intubated for >72 hours. Note: in the event of extubation and re-intubation, the calculation for the number of hours the subject has been intubated begins at the first intubation
* Require or anticipated need for extracorporeal membrane oxygenation (ECMO) Suspected or proven septic shock or shock ;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is >5 times higher than the upper limit normal range;
* Severe chronic respiratory disease (e.g., known chronic obstructive pulmonary disease [COPD], pulmonary arterial hypertension [PAH], idiopathic pulmonary fibrosis [IPF], interstitial lung disease [ILD]) requiring supplemental oxygen therapy or mechanical ventilation pre-hospitalization (e.g., prior to COVID-19 diagnosis)
* Use of prohibited medications
* Participants with severe COVID-19 who received convalescent plasma or COVID-19 vaccine , or anti-spike (S) SARS-CoV-2 therapy.
* Moribund condition in the opinion of the clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2021-02-25 (Estimated); Primary Completion 2021-05-25 (Estimated); Study Completion 2021-11-25 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate at D29 | Day 29
  The mortality rates in placebo and treatment groups regardless of the cause of death.

SECONDARY OUTCOMES:
All-cause mortality rate at Day 60 | Day 60
  The mortality rates in placebo and treatment groups regardless of the cause of death.
Time to discontinue mechanical ventilation (MV) at Day 29 | Baseline through Day 29
  The number of days from randomization to discontinue MV support
Time to improvement of two categories on WHO 10-Point Ordinal Scale from baseline at Day 29 | Baseline through Day 29
  The number of days from baseline to two categories decreases on World Health Organization (WHO) 10-Point Ordinal Scale at Day 29.
Time to discontinue supplemental oxygen at Day 29 | Baseline through Day 29
  The number of days from randomization to discontinue supplemental oxygen support
Time to hospital free at Day 29 | Baseline through Day 29
  The number of days from randomization to subject's discharge from hospital.
Change from baseline in viral shedding as measured by quantitative reverse transcription polymerase chain reaction (RT-qPCR) | Baseline through Day 29
  Change from baseline in viral shedding
SAE | Day 1 through Day 120
  SAEs collected from Day 1 to Day 120
Anti-drug antibody (ADA) | Day 29, Day 120
  ADA will be tested at Day 29 and Day120 after SCTA01/placebo administration

CONTACTS AND LOCATIONS:
Overall Officials: Zhanghua Lan, PhD, Study Director — SCT

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343